CLINICAL TRIAL: NCT04009603
Title: Comparison of Probiotics, Metformin and Their Combination Therapy in Improving Symptoms of Polycystic Ovarian Syndrome.̎- A Randomized Clinical Trial
Brief Title: Comparison of Probiotics, Metformin & Their Combination Therapy in the Treatment of PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr. Urooj Zafar, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 651118UZPHA
Record Dates: First submitted 2019-03-28; First posted 2019-07-05 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metformin (Active Comparator): Group no 1(26 patients) Metformin tablets at a dose of 500mg BD for 12 weeks
  Interventions: Drug: Metformin
- Probiotic (Experimental): Group no 2(26 patients): will be given probiotics alone at a dose of 180mg B.D for 12 weeks
  Interventions: Drug: Probiotic Agent
- Metformin and Probiotic (Experimental): Group no 3(26 patients): will be given metformin 500mg B.D and probiotics 180mgram O.D. for 12 week
  Interventions: Drug: Probiotic Agent; Drug: Metformin

INTERVENTIONS:
Drug: Probiotic Agent — Probiotics are live microorganisms, which when administered in adequate amounts confer a health benefit effects on the host.
  Many clinical trials have been done on probiotic which show its use as a single or as an adjuvant drug therapy for various diseases with no or rare side effects. It is now frequently used agent for various diseases.
  Apart from this many studies have been published related to effects of probiotics on PCOS, which shows effectiveness of probiotics when used for 8 to 12 weeks with no adverse effects observed by these micro-organisms but none of the study have compare it with standarad drug
  Other Names: Ecotec
  Arms: Metformin and Probiotic; Probiotic
Drug: Metformin — Metformin, an insulin sensitizer, is an oral biguanide that is most commonly prescribed for the management of type II diabetes mellitus and various symptoms of PCOS. It is derived from the extract of Galega officinalis.
  It remediates hyperglycemia through activation of AMPK which stimulates glucose uptake and its consumption; promote fatty acid oxidation along with suppression of hepatic glucose production. It is also involved in increase GLUT4 translocation in the muscle and fat leading to decrease hepatic lipid synthesis. Moreover, It is also reported that it decreases gut absorption of glucose by increasing the glucagon-like peptide-1 (GLP-1) in this way, it reduces the insulin requirement too.All of these actions of metformin decrease insulin resistance and thus improve the state of hyperinsulinemia associated with diabetes and PCOS
  Other Names: glucophage
  Arms: Metformin; Metformin and Probiotic

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common gynecological state worldwide characterized by numerous small cysts in the ovaries mainly due to the imbalance of endocrine hormones in premenopausal women. Metformin is long being used for different symptoms of PCOS along with other medication. This study involves the assessment of different parameters of PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a hormonal disorder affecting the women of reproductive age. It is a heterogeneous health condition that affects 1 in every 10 women of childbearing age. Women of all races and ethnicities are at risk for PCOS, but risk increases multiple folds if the BMI is greater than 30kg/m2. The common signs and symptoms, the women usually represent with are menstrual irregularities, hyperandrogenemia and multiple cysts in ovaries. The exact cause of PCOS is still unknown but genetic and obesity is considered to be the most common cause.

Metformin has been considered as the first line agent for the treatment of non-insulin dependent diabetes mellitus and up till now it has been used as a first line drug for PCOS. Despite its beneficial effects in PCOS it has several adverse effects. Moreover, patients usually seek two or more drugs along with metformin to relieve maximum symptoms of PCOS like for ovulation clomiphene citrate must be given etc. So there is a need of novel and comprehensive agent that can prove to be effective in improving maximum symptoms of this disease. Probiotics have received renewed attention in the 21st century through research studies. World Health Organization's (WHO) 2001 defines probiotics as live micro-organisms that, when administered in adequate amounts, confer a health benefit on the host. In recent year it has shown tremendous promising effect in treatment of different diseases like diarrhea, gingivitis and obesity etc with negligible side effects.

In this context the investigators are going to evaluate and compare the effects of probiotics, metformin and their combination therapy in treatment of various symptoms of PCOS.60 newly diagnosed PCOS patient will be assigned in the open label randomized clinical trial. As mentioned above patients will be divided into three groups with 20 patients each. In group 1, the dosage of metformin will be 500mg B.D and 2 gm of probiotic sachet O.D, the second group will be given metformin 500mg B.D. and the third group will be 2mg of probiotics B.D. It would be a follow-up study that would be conducted in Gynecology OPD of Tertiary Care Hospital

ELIGIBILITY:
Inclusion Criteria:

* The patient will be included according to the Rotterdam European Society for Human Reproduction and Embryology/American Society for Reproductive Medicine sponsored a PCOS consensus criterion which says the presence of any two of the following three features must be present for the patient to be diagnosed as a case of PCOS:

  * Oligomenorrhea and/or amenorrhea (Oligomenorrhea>45 days or <8 cycles per year and amenorrhea >3 months in women with previous periodic menses) for a period of 6 months
  * Clinical and/or biochemical hyperandrogenemia, the presence of acne, hirsutism (FG score>8), and alopecia
  * Polycystic ovaries on sonography (>12 follicles in one or both ovaries, 2-9 mm in diameter and/or increased ovarian volume >10 mL).

Exclusion Criteria:

* History of chronic diseases
* Allergic to probiotic or metformin
* Current or previous (within the last 6 months) use of chemotherapy or other drugs.
* History of smoking
* Individuals with autoimmune disease
* Individuals with autoimmune disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Biochemical parameter: | 12 weeks
  Fasting serum glucose:
  The blood sample for FBS will be collected on day 2 or 3 of the menses. The blood samples will be taken before the start and at the end of the treatment.
  fasting glucose 80-100 mg/dl
Hormonal parameter: | 12 weeks
  Androgens:
  The concentration of these hormones will be evaluated at the baseline and at the end of treatment usually in the morning between 8:00 am to 9:00 am after overnight fasting
  Serum testosterone:15 and 70 ng/dL
Change in cyst size on Ultrasonography | 12 weeks
  Ovary cyst size:
  The size of the cyst will be measured before the start and at the end of the study, considering 12 or more follicles in at least 1 ovary or both-measuring 2-9 mm in diameter-or a total ovarian volume greater than 10 cm3
Luteinizing Hormone | 12 weeks
  LH
  The concentration of this endocrine hormones is determined will be obtained on day 2 or 3 of the normal menstruation cycle and at any time in women with amenorrhea.
  LH: 1.9 to 12.5 IU/L
INSULIN LEVELS | 12 weeks
  Fasting serum insulin:
  The sample is collected after fasting of 12 to 14 hours will be measured before and after intervention
  fasting insulin < 25 mIU/L
Lipid | 12 weeks
  Lipid profile:
  1. Total cholesterol
  2. LDL
  3. HDL
  4. Triglyceride
  The serum lipid concentrations will be evaluated spectrophotometrically by means of commercial kits at baseline and at the end of the study
  Total cholesterol < 200
  Triglyceride: <150 mg/dl
  HDL: > 60mg/ dl
  LDL: < 130mg /dl
Follicle-stimulating hormone | 12 weeks
  The concentration of this endocrine hormones is determined will be obtained on day 2 or 3 of the normal menstruation cycle and at any time in women with amenorrhea.
  LH: 4.5 to 21.5 IU/L
LH and FSH ratio | 12 weeks
  LH:FSH The serum levels of FSH:LH ratio will be assessed before the start and at the end of the management on day 2 or 3 of the normal menses and at any time in women with amenorrhea.
  1.5:1

SECONDARY OUTCOMES:
Change in Physical symptoms in PCOS | 12 weeks
  Weight:
  The body weight of the females will be recorded at baseline and at the end of the treatment with the help of weighing machine in kg.
Menstruration | 12 weeks
  Menstrurational irregularities:
  All study participants will be asked about menstruation irregularities at the time of enrollment.They will also be enquired about for long they have their cycles have been disturbed.They will be asked to maintain their cycle dates as well.
Hirsutism | 12 week
  Hirsutism:
  History and physical examination, including pelvic examination at the start and at the end of treatment using the Ferriman-Gallwey scale for hirsutism.
Acne | 12 week
  Acne:
  Acne score will be taken at baseline and at the end of the treatment through the Global Acne grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Urooj Zafar, M.Phil, Principal Investigator — Ziauddin University
Locations (1):
- Dr. Urooj, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahmadi S, Jamilian M, Karamali M, Tajabadi-Ebrahimi M, Jafari P, Taghizadeh M, Memarzadeh MR, Asemi Z. Probiotic supplementation and the effects on weight loss, glycaemia and lipid profiles in women with polycystic ovary syndrome: a randomized, double-blind, placebo-controlled trial. Hum Fertil (Camb). 2017 Dec;20(4):254-261. doi: 10.1080/14647273.2017.1283446. Epub 2017 Feb 1. PMID 28142296
- [Result] Shoaei T, Heidari-Beni M, Tehrani HG, Feizi A, Esmaillzadeh A, Askari G. Effects of Probiotic Supplementation on Pancreatic beta-cell Function and C-reactive Protein in Women with Polycystic Ovary Syndrome: A Randomized Double-blind Placebo-controlled Clinical Trial. Int J Prev Med. 2015 Mar 24;6:27. doi: 10.4103/2008-7802.153866. eCollection 2015. PMID 25949777
- [Result] Karamali M, Eghbalpour S, Rajabi S, Jamilian M, Bahmani F, Tajabadi-Ebrahimi M, Keneshlou F, Mirhashemi SM, Chamani M, Hashem Gelougerdi S, Asemi Z. Effects of Probiotic Supplementation on Hormonal Profiles, Biomarkers of Inflammation and Oxidative Stress in Women With Polycystic Ovary Syndrome: A Randomized, Double-Blind, Placebo-Controlled Trial. Arch Iran Med. 2018 Jan 1;21(1):1-7. PMID 29664663
- [Result] Liao D, Zhong C, Li C, Mo L, Liu Y. Meta-analysis of the effects of probiotic supplementation on glycemia, lipidic profiles, weight loss and C-reactive protein in women with polycystic ovarian syndrome. Minerva Med. 2018 Dec;109(6):479-487. doi: 10.23736/S0026-4806.18.05728-2. Epub 2018 Sep 24. PMID 30256077
- See also: Effects of Probiotic Supplementation on Pancreatic β-cell Function and C-reactive Protein in Women with Polycystic Ovary Syndrome: A Randomized Double-blind Placebo-controlled Clinical Tria — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4387688/
- See also: Meta-analysis of the effects of probiotic supplementation on glycemia, lipidic profiles, weight loss and C-reactive protein in women with polycystic ovarian syndrome. — https://europepmc.org/abstract/med/30256077